CLINICAL TRIAL: NCT04134910
Title: The Role of Disc Nutrition in the Etiology and Clinical Treatment of Disc Degeneration
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Grants funds ended/spent out on other aims prior to being able to being this study
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B3118-W
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Back Pain; Intervertebral Disc Degeneration
Keywords: spine; intervertebral disc; physical therapy; imaging
MeSH Terms: conditions — Back Pain; Intervertebral Disc Degeneration | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Physical therapy (Experimental): Subjects will be prescribed a 6-week physical therapy regimen consisting of one 45 minute in office visit per week, and home exercises performed daily. The in-office visits with a physical therapy provider will consist of the application of manual therapy, particularly high-velocity, low amplitude thrust mobilization in the anterior/posterior direction of the lumbar spine. In office visits will also include supervised repeated motion of the lumbar spine into extension (McKenzie therapy, 3 sets of 10 repetitions, in prone and standing positions) Patients will be instructed to complete these repeated extension exercises at home daily for the 6 week period.
  Interventions: Procedure: Physical Therapy

INTERVENTIONS:
Procedure: Physical Therapy — Subjects will be prescribed a 6-week physical therapy regimen consisting of one 45 minute in office visit per week, and home exercises performed daily. The in-office visits with a physical therapy provider will consist of the application of manual therapy, particularly high-velocity, low amplitude thrust mobilization in the anterior/posterior direction of the lumbar spine. In office visits will also include supervised repeated motion of the lumbar spine into extension (McKenzie therapy, 3 sets of 10 repetitions, in prone and standing positions) Patients will be instructed to complete these repeated extension exercises at home daily for the 6 week period.

SUMMARY:
The purpose of this research study is to examine the effects of physical therapy on the spinal discs. Back pain is the number one cause of disability in the US, and the spine is the most common location of chronic pain in Veterans. Physical therapy is often very effective at improving patients' back pain, but it does not work for everyone, and it is not understood how physical therapy alters the tissues within the spine. With this research the investigators hope to learn if the investigative team can measure changes to the spinal discs on MRI scans that might predict if a patient's back pain will improve with physical therapy or not.

DETAILED DESCRIPTION:
Low back pain, which is frequently associated with intervertebral disc degeneration, is the most common cause of adult disability in the United States. Among active service members, the incidence of disc degeneration more than doubled from 2001 to 2010, with over 68,000 days of lost duty time attributed to disc degeneration.2 The most common location of chronic pain in Veterans is the spine. The incidence of back pain in the general public has remained relatively stable over the past decade, however, there has been more than a 50% increase in the number of Veterans diagnosed with back pain. The intervertebral discs are the largest avascular structures in the body, and therefore cells within the disc rely on transport from the small vessels in the adjacent vertebral endplate to receive nutrients and expel waste products. Despite the immense social and economic burden of back pain, the etiology of disc degeneration remains poorly understood. Because of the avascular nature of the disc, it has been speculated that poor disc nutrition characterized by reduced trans-endplate transport into the disc could contribute to the initiation and progression of degeneration. If a reduction in trans-endplate transport of nutrients and waste products is a primary contributor to the initiation and progression of the degenerative cascade, then enhancing disc nutrition may have a therapeutic effect. Physical therapy and exercise can be very effective in managing back pain for certain patients, yet it is not fully understood why certain patients respond to physical therapy and others do not, and what effects such interventions have on disc nutrition and disc health. The goal of this study is to undertake a pilot study to determine the feasibility and preliminary outcomes of utilizing quantitative MRI in human patients to quantify changes in disc health and trans-endplate transport over the course of physical therapy.

To do so, patients with low back pain and concomitant disc degeneration, who have not had prior spinal surgery, will be recruited. Recruited patients will undergo MRI T2-mapping and post-contrast enhanced T1-mapping of their lumbar spines at 1.5T to measure disc health and nutrition, respectively. Patients will then begin a 6 week physical therapy treatment regimen, after which the same MRI scans will be performed again on each patient. Pain and disability level of patients will be assessed via the visual analog scale (VAS) and Oswestry Disability Index (ODI) questionnaires, both pre- and post-treatment. Lumbar active range of motion will also be quantified at the initial and final in-office physical therapy session. Inclinometers will be placed at the thoracolumbar junction and sacrum, and the patient asked to bend forward and backward. Lumbar flexion will be quantified as the difference in motion between the two inclinometers.

Significant differences T1 and T2 values in the disc, as well as VAS and ODI scores and lumbar range of motion, before and after physical therapy will be assessed via a paired t-test, with significance defined as p<0.05. Univariate linear correlations between the changes in T1 or T2 values and changes in VAS, ODI scores and lumbar range of motion will be performed to determine if altered disc health or nutrition with physical therapy is significantly correlated with improvements in pain and disability.

ELIGIBILITY:
Inclusion Criteria:

* Current activity limiting low back pain
* With symptoms of any duration
* With or without symptoms extending distal to the buttocks
* Medically stable
* Candidate for physical therapy

Exclusion Criteria:

* Documented history of prior spinal surgery
* Contraindications to MRI including:

  * claustrophobia
  * pregnancy
  * implanted electronic devices

    * pacemakers, cochlear implant, insulin pumps, etc
  * metallic foreign bodies

    * i.e. shrapnel
  * documented history of contraindications to gadodiamide (Omniscan) administration:

    * chronic severe kidney disease
    * acute kidney injury
    * impaired elimination of gadolinium based contrast agents
    * pre-existing renal insufficiency
    * a prior hypersensitivity reaction to MRI contrast

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Change in Disc T2 relaxation time | 0 to 6 weeks
  Subjects will undergo MRI scanning to obtain T2-maps of the lumbar spine before and after 6 weeks of physical therapy. T2 relaxation times of the disc tissues are calculated from the images.
Change in Visual Analog Scale (VAS) score | 0 to 6 weeks
  Subjects will complete a visual analog scale (VAS) for their back pain before and after 6 weeks of physical therapy. This is a scale from 0 (no pain) to 15 (the worst imaginable pain).
Change in Lumbar Range of Motion | 0 to 6 weeks
  Lumbar range of motion will be measured using inclinometers placed on the subject's upper and lower back, at both the index and final in-office physical therapy visit.
Change in Disc T1 relaxation time | 0 to 6 weeks
  Subjects will undergo MRI scanning to obtain post-contrast enhanced T1 maps of the lumbar spine before and after 6 weeks of physical therapy. To obtain the T1 maps, an intravenous catheter will be placed, and 0.1 mmols/kg of Omniscan will be administered. T1 MRIs will be acquired prior to and 2 hours following Omniscan administration. T1 relaxation times of the disc tissues are calculated from the images.
Change in Oswestry Disability Index (ODI) score | 0 to 6 weeks
  Subjects will complete the ODI questionnaire before and after 6 weeks of physical therapy. This is a scale from 0 (no disability) to 50 (bed bound).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E. Gullbrand, PhD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (1):
- Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No